CLINICAL TRIAL: NCT00086320
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study With an Open-label Extension Evaluating Paliperidone Extended Release Tablets in the Prevention of Recurrence in Subjects With Schizophrenia
Brief Title: A Study of Effectiveness and Safety of Paliperidone Extended-release (ER) Tablets in the Prevention of Recurrence in Adult Patients With Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004384
Record Dates: First submitted 2004-06-30; First posted 2004-07-01 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; paliperidone; Risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to determine the efficacy (effectiveness) and safety of paliperidone ER compared with placebo in the prevention of recurrence of symptoms of schizophrenia.

DETAILED DESCRIPTION:
Paliperidone ER is currently being investigated as treatment for the acute symptoms of schizophrenia and also as maintenance treatment. This trial is designed to evaluate efficacy and safety of paliperidone ER in prevention of recurrence of psychotic symptoms in patients with schizophrenia. This trial is a randomized (patients will be assigned to different treatment groups based solely on chance), double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), placebo-controlled, parallel-group, multicenter study consisting of 5 phases: a screening phase of up to 5 days; a 8-week open-label run-in phase, during which all patients will be treated with open-label, flexibly dosed paliperidone ER (3 to 15 mg) orally once daily to identify a dose that will achieve control of their acute psychotic symptoms (only patients who maintain a stable dosage regimen and have a total Positive and Negative Syndrome Scale [PANSS] score </=70; Clinical Global Impression Scale - Severity [CGI-S] </=4; and scores of </=4 for PANSS items for delusions, conceptual disorganization, hallucinatory behavior, suspiciousness/persecution, hostility, and uncooperativeness during the last 2 weeks of the run-in phase will be eligible to continue in the stabilization phase); a 6-week open-label stabilization phase, patients who maintain control of their acute psychotic symptoms at the paliperidone ER dosage identified during the run-in phase and meet the total PANSS score, CGI-S, and PANSS items scores throughout the stabilization phase will be randomized to receive either flexibly dosed paliperidone ER, starting at the dose maintained during the stabilization phase of the study, or placebo; a double-blind treatment phase of variable duration, during which patients will be followed until they meet either defined criteria for recurrence or the study ends; a 52-week open-label extension phase for patients who experience a recurrence event during the double-blind phase of the study, or who remain recurrence free for the entire double-blind phase of the study. Efficacy will be assessed using the PANSS and CGI-S scores that will be collected every week, every 2 weeks, or every 4 weeks throughout. Safety assessments include the incidence of adverse events throughout the study; measurement of vital signs (orthostatic pulse rate, orthostatic blood pressure, and temperature); and clinical laboratory tests. In the run-in, double-blind, and open-label extension phases of the study, paliperidone ER or matching placebo will be flexibly dosed in the range 3 to 15 mg orally once a day (3, 6, 9, 12, or 15 mg/day). The dosage in the stabilization phase will be fixed throughout at the dosage that achieved symptom control in the run-in phase.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia at least 1 year before screening
* experiencing an acute schizophrenic episode with a total PANSS score between 70 and 120
* agree to be hospitalized for a minimum of 14 days at the start of the study
* capable of administering study medication themselves or have assistance with study medication administration consistently available throughout the study
* resided at the same address continuously for at least 30 days prior to screening
* able and willing to fill out self administered questionnaires
* washout of antiparkinsonian medications, beta-blockers
* antiepileptics, lithium 3 days prior to the start of the run-in phase

Exclusion Criteria:

* DSM-IV Axis I diagnosis other than schizophrenia
* DSM-IV diagnosis of substance dependence within 6 months prior to screening (nicotine and caffeine dependence are not exclusionary)
* preexisting severe gastrointestinal narrowing (pathologic or iatrogenic)
* injection of a depot antipsychotic within 120 days before screening, or use of paliperidone palmitate within 10 months before screening
* previous history of lack of response to risperidone when acutely psychotic
* history of neuroleptic malignant syndrome
* significant risk of suicidal or violent behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2004-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Time to recurrence, defined as the time between randomization to treatment in the double-blind period and the first documentation of a recurrence.

SECONDARY OUTCOMES:
Change in PANSS total and subscale scores from randomization to each visit and to the end of the study. Change from baseline in CGI-S at each assessment time point and at endpoint. Incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Mathews M, Gopal S, Singh A, Nuamah I, Pungor K, Tan W, Soares B, Kim E, Savitz AJ. Comparison of Relapse Prevention with 3 Different Paliperidone Formulations in Patients with Schizophrenia Continuing versus Discontinuing Active Antipsychotic Treatment: A Post-Hoc Analysis of 3 Similarly Designed Randomized Studies. Neuropsychiatr Dis Treat. 2020 Jun 19;16:1533-1542. doi: 10.2147/NDT.S221242. eCollection 2020. PMID 32606705
- [Derived] Weiden PJ, Kim E, Bermak J, Turkoz I, Gopal S, Berwaerts J. Does Half-Life Matter After Antipsychotic Discontinuation? A Relapse Comparison in Schizophrenia With 3 Different Formulations of Paliperidone. J Clin Psychiatry. 2017 Jul;78(7):e813-e820. doi: 10.4088/JCP.16m11308. PMID 28640988
- [Derived] Kramer M, Simpson G, Maciulis V, Kushner S, Vijapurkar U, Lim P, Eerdekens M. Paliperidone extended-release tablets for prevention of symptom recurrence in patients with schizophrenia: a randomized, double-blind, placebo-controlled study. J Clin Psychopharmacol. 2007 Feb;27(1):6-14. doi: 10.1097/JCP.0b013e31802dda4a. PMID 17224706
- See also: A Study of Effectiveness and Safety of Paliperidone Extended-Release (ER) Tablets in the Prevention of Recurrence in Adult Patients With Schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=587&filename=CR004384_CSR.pdf